CLINICAL TRIAL: NCT06298799
Title: RETRO-PROSPECTIVE OPEN STUDY TO ASSES GENETIC VARIABILITY AS A BASIS FOR PREDICTION OF THE RESPONSE TO GLP1 TREATMENT
Brief Title: GENETIC VARIABILITY TO GLP1 TREATMENT
Acronym: GLP1 treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GENGE (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GEN-GE-001-IL
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Sequence Analysis, DNA; Base Sequence

STUDY DESIGN:
Intervention Model Description: The study population consists of two cohorts:
  A. Type 2 Diabetic participants cohort B. Healthy participants cohort
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of DNA/RNA samples (Other): Type 2 Diabetic participants cohort or Healthy participants cohort who will perform Collection of DNA/RNA samples
  Interventions: Genetic: DNA Sequencing and Analysis; Genetic: differential expression analysis with RNA-sequencing (RNA seq) experiments

INTERVENTIONS:
Genetic: DNA Sequencing and Analysis — DNA extracted from saliva / oral mucosa will be tested for diversities reported in the literature known to be associated with T2DM and Obesity and which may have a potential impact on the response to treatment with Semaglutide. In addition, the DNA will be screened for new diversities that have a potential impact on the response to treatment. working assumption of the study is that there can be 3 types of genetic variants that affect the drug's effectiveness and/or side effects.
Genetic: differential expression analysis with RNA-sequencing (RNA seq) experiments — Performing small RNA sequencing experiments on an Illumina Next-Generation Sequencing (NGS) machine to investigate microRNAs (miRNAs) or other small non-coding RNAs involves specific steps tailored to the unique characteristics of these molecules

SUMMARY:
The goal of this retrospective study is to assess whether a selection of genetic variants may allow us to identify individuals who will have a satisfactory response after GLP-1 treatment in terms of weight loss, sugar level reduction, and adverse events.

Participants will The study consists of a single visit at the diabetes unit clinic at the involved study sites. The following will be performed for every subject at the study screening enrollment visit:

* Informed consent
* Study eligibility (Inclusion / Exclusion criteria)
* Collection of demographic data (age (date of birth), gender, ethnic origin)
* General and T2DM medical history review (per subject file)
* Concomitant medication review (at enrollment)
* Physical attributes (Body Weight, Height, BMI)
* Allocation to study cohort and study subgroup
* Saliva and blood collection for genetic tests
* Self-reported questionnaire for Ozempic (Semaglutide) experience

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes (for participant in Cohort A) or Obese (for participant in Cohort B) and treated with Ozempic (Semaglutide) S.C. injection for at least 24 weeks.
2. Subject is male/female between 18 to 80 years old (both inclusive) at the time of enrollment.
3. Subject BMI above 30 kg/m2 at treatment initiation.
4. Subject does not belong to any vulnerable population, is willing and able to provide written informed consent prior to any study procedure.
5. Participant understands the nature of the procedure and is willing and able to comply with all requirement of the protocol.

Exclusion Criteria:

1. Subject falls under contraindications to Ozempic (Semaglutide) label
2. Subject known or suspected for hypersensitivity to any GLP-1RA or related products, or allergic constitution
3. Subjects suffers from any other condition affecting body weight.
4. Subject with history of chronic or acute pancreatitis
5. Subject have a history of a major cardiovascular and/or cerebrovascular disease within the 6 months before screening.
6. Presence or history of malignant neoplasm within 5 years prior to screening day.
7. Subject suffers from any renal impairment (Cr > 2 mg/dl).
8. Subject suffers from any impaired hepatic function (ALT, AST or GGT 2-fold higher than normal upper limit).
9. Any disorder, which in the investigator's opinion might jeopardize patient's safety or compliance with the protocol.
10. Subject is a female who is pregnant, breastfeeding or intends to become pregnant or is of child bearing potential without medically acceptable methods of contraception.
11. Participation in another clinical study in prior 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetic variants and miRNA expressions associated with changes in BMI. | 12 months
  Identify genetic variants and miRNA expressions that affects the response to GLP-1 treatment associated with changes in BMI.

SECONDARY OUTCOMES:
Genetic variants and miRNA expressions associated with changes in A1c. | 12 months
  Identify genetic variants and miRNA expressions that affects the response to GLP-1 treatment associated with changes in A1c.

OTHER OUTCOMES:
Genetic variants and miRNA expressions associated with side effects. | 12 months
  Identify genetic variants and miRNA expressions that affects the response to GLP-1 treatment associated with side effects.
Demographic parameters that affect GLP1 AG therapy. | 12 months
  To identify demographic parameters that affect the response to GLP1 AG therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambem medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No